CLINICAL TRIAL: NCT07196111
Title: Evaluation of the Safety and Efficacy of BAFFR CAR-T Therapy in Clinical Studies for Recurrent/Refractory B Cell Tumors.
Brief Title: BAFFR CAR-T Treatment for Relapsed/Refractory B-cell Tumors
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangzhou Bio-gene Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YD-003
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: B Acute Lymphoblastic Leukemia/Lymphoma
Keywords: BAFFR
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAFFR CAR-T cell injection (Experimental): Dose escalation: Three dose levels were designed, and if the maximum tolerated dose (MTD) was not found at the highest level, no further dose escalation was to be performed. Approximately 12-18 subjects were planned to be enrolled in the dose-escalation phase to evaluate the safety and tolerability of BAFFR CAR-T injection and to determine the MTD and/or the recommended phase II dose (RP2D). Dose Expansion: During or after the dose escalation process, if a certain dose group is determined to have preliminary anti-tumor effects and controllable safety, it can be extended at this dose level to further evaluate the tolerance and safety of BAFFR CAR-T injection, and to preliminarily evaluate its effectiveness.
  Interventions: Biological: BAFFR CAR-T

INTERVENTIONS:
Biological: BAFFR CAR-T — A single infusion of BAFFR CAR-T Injection administered intravenously.

SUMMARY:
This study is a single-arm, multicenter clinical trial of dose escalation and dose expansion.

DETAILED DESCRIPTION:
This study is a single-arm, mult-center clinical trial of dose escalation and dose expansion, primarily aimed at evaluating the safety, tolerability, and preliminary efficacy of BAFFR CAR-T cell infusion in subjects with relapsed/refractory B-cell tumors.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or their guardian understands and voluntarily signs the informed consent form and expects to complete the follow-up examinations and treatments of the research protocol；
2. Age 18-85 years old (inclusive), gender unrestricted;
3. The definition of refractory in patients with B-cell lymphoma is as follows:

   * no response to the most recent treatment, including:

     1. the best response to the most recent treatment regimen is disease progression (PD);
     2. or the best response to the most recent treatment is stable disease (SD) and the duration does not exceed 6 months after the last administration;
   * or unsuitable or unwilling to undergo autologous hematopoietic stem cell transplantation (ASCT), or ASCT refractory, including:

     1. disease progression or recurrence within ≤ 12 months after ASCT;
     2. or if salvage treatment is administered after ASCT, the subject must have no response or relapse after the last treatment;
4. B-ALL/LBL patients, refractory definition: failure to achieve complete remission (bone marrow blast cells ≥ 5% or persistence of extramedullary lesions) after standard induction or salvage therapy, or early relapse (<12 months) after remission with no response to re-induction therapy.
5. Patients with relapsed/refractory acute B-cell lymphoma who have previously been treated with anti-CD20 targeted agents (unless documented as CD20 negative) and anthracycline agents;
6. Patients with lymphoma must have at least one measurable lesion from baseline according to the revised IWG criteria for assessing the efficacy of malignant lymphoma；
7. The organ functions well；
8. ECOG performance status score 0-3 and estimated survival time greater than 3 months.

Exclusion Criteria:

1. Have other malignant tumors within 3 years before screening, excluding adequately treated cervical carcinoma in situ, papillary thyroid carcinoma, basal cell or squamous cell skin cancer, local prostate cancer after radical prostatectomy, and ductal carcinoma in situ after radical prostatectomy.
2. Hepatitis B surface antigen (HBsAg) positive, hepatitis B core antibody (HBcAb) positive and peripheral blood HBV-DNA higher than the detection limit; Hepatitis C virus (HCV) antibody positive; Persons with human immunodeficiency virus (HIV) antibody positive; Cytomegalovirus (CMV) DNA positive cases; EBV-DNA positive patients; The syphilis antibody was positive.
3. Those with a history of anaphylaxis [A history of anaphylaxis was defined as an allergic reaction of grade 2 or higher, in which any of the following clinical manifestations occurred: Airway obstruction (rhinorrhea, cough, stridor, dyspnea), Tachycardia, Hypotension, Arrhythmia, Gastrointestinal symptoms (nausea, vomiting), Incontinence, Laryngeal edema, Bronchospasm, Cyanosis, Shock, Respiratory, cardiac arrest] or known to be allergic to any of the drug active ingredients, excipents, or mouse-derived products or xenoproteins included in this trial (including the lymphatic cells clearance protocol).
4. Have severe cardiac disease, including but not limited to severe arrhythmia, unstable angina, massive myocardial infarction, New York Heart Association class III or IV cardiac dysfunction, and refractory hypertension.
5. Previous organ transplantation or preparation for organ transplantation (excluding hematopoietic stem cell transplantation).
6. Active autoimmune or inflammatory diseases (e.g., Guillain-Barre syndrome (GBS), amyotrophic lateral sclerosis (ALS)) and clinically significant active cerebrovascular diseases (e.g., cerebral edema, posterior reversible encephalopathy syndrome (PRES)).
7. Patients with cancer emergencies (such as spinal cord compression, intestinal obstruction, leukostasis, tumor lysis syndrome, etc.) requiring emergency treatment before screening or reinfusion.
8. Presence of uncontrolled bacterial, fungal, viral, or other infection requiring antibiotic treatment.
9. Patients who had undergone major surgery (excluding diagnostic surgery and biopsy) within 4 weeks before lymphatic cells clearance or planned to undergo major surgery during the study period, or who had not fully healed the surgical wound before enrollment.
10. Persons with severe mental illness.
11. Within 1 week before the collection of peripheral blood mononuclear cells (PBMC), patients who use granulocyte colony-stimulating factor (G-CSF), granulocyte macrophage colony-stimulating factor (GM-CSF) and other hematopoietic cytokine drugs that have an impact on the patient's blood picture (if it is a long-acting preparation, it is 2 weeks) and have an impact on cell preparation as judged by the investigator .
12. Within 2 weeks before PBMC collection, patients were receiving hormonal or immunosuppressive drugs that were judged by the investigator to have an effect on cell production.

    1. hormone: subjects who were receiving systemic steroid therapy within 2 weeks before PBMC collection and who required long-term systemic steroid therapy (except inhaled or topical use) as judged by the investigator during the treatment.
    2. Immunosuppressive agents: those who were receiving immunosuppressive agents within 2 weeks before PBMC collection.
13. Vaccination with live (attenuated) virus vaccine within 4 weeks prior to screening.
14. Alcoholics or those with a history of substance abuse.
15. Patients who, in the investigator's judgment and/or clinical criteria, have contraindications to any study procedure or other medical conditions that may put them at unacceptable risk.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2028-10-09 (Estimated); Study Completion 2028-12-09 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity Rate | Up to 28 days after CAR-T infusion.
  After the infusion of CAR-T, subjects still experienced adverse events, meeting the DLT definition, related to or possibly related to CAR-T infusion after optimal supportive treatment.
Incidence of Treatment-Emergent Adverse Events | Up to 24 months.
  Count the Incidence of adverse events.

SECONDARY OUTCOMES:
Concentration of CAR-T cells after Infusion (PK) | Up to 24 months.
  CAR-T in peripheral blood after infusion
overall response rate, ORR | Up to 24 months.
  Defined as the proportion of subjects achieving complete response(CR), complete remission with incomplete blood cell recovery (CRi), or partial response(PR).
Concentration of Cytokine after Infusion (PD) | Up to 24 months.
  Calculate the change of cytokine concentration in peripheral blood after After CAR-T infusion. Cytokines include IL-2、IL-6 and so on.